CLINICAL TRIAL: NCT05587764
Title: A Post Market Clinical Follow-up Study to Evaluate the Safety and Clinical Performance of the Tempus Pro, a Multi-parameter Vital Signs Monitoring Device With Specific Reference to ECG Recordings and Data Transmission Using Telemedicine
Brief Title: Tempus Pro Monitor Registry
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: North American Science Associates, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCTCRDTTempusProRegi20211168
Record Dates: First submitted 2022-10-13; First posted 2022-10-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Sudden Cardiac Arrest; Emergency Care
Keywords: Tempus Pro; IntelliSpace Corsium
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Standard of Care: Standard of Care for emergency care
  Interventions: Diagnostic Test: Standard of Care

INTERVENTIONS:
Diagnostic Test: Standard of Care — Standard of care for emergency events per local guidelines.

SUMMARY:
A multicenter, prospective and retrospective, observational, post market study.

DETAILED DESCRIPTION:
This observational study is to collect real-world data on the safety and performance of the Tempus Pro device, its accessories and the IntelliSpace Corsium telemedicine software device when used according to its intended purpose and the instructions for use, when used for patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

Patients monitored by using Tempus Pro during pre-hospital care (ambulance transportation)

One or more 12-lead ECG recorded

Use of 3 or more of the following sensors to measure vital signs

* NIBP (Non-Invasive Blood Pressure)
* HR (Heart Rate)
* SpO2 (Oxygen Saturation)
* PVI (Pleth Variability Index)
* SpCO (Carboxyhemoglobin)
* SpOC (Oxygen Content)
* SpHb (Total Hemoglobin)
* SpMet (Methemoglobin Saturation)
* EtCO2 (End-tidal Carbon Dioxide)

Exclusion Criteria:

* None defined

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pre- and inter-hospital transfer: emergency patients (adults and pediatrics).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Clinician assessment of 12-lead ECG reports | through study completion, an average of 1 year
  The proportion of 12-lead ECG pairs that are identical, after a cardiologist's review of printouts from Corsium IntelliSpace (transmitted) ECG and the original ECG from the Tempus Pro device.
Diagnostic quality of 12-lead | through study completion, an average of 1 year
  The printed patient record ECG will be independently reviewed for abnormalities and distortion by a clinician. The clinician will note any abnormalities altering diagnostic quality.
Consistency of transmitted vital signs by Tempus Pro via IntelliSpace Corsium | through study completion, an average of 1 year
  The number and proportion of patient vital sign data points, comparing direct data with identical units of measure from printouts from IntelliSpace Corsium (transmitted) vital signs and the original vital signs from the Tempus Pro device.

SECONDARY OUTCOMES:
Number of all activated alarms | through study completion, an average of 1 year
  The 'Summary Record of Care' indicates all alarms - for all alarm-settable parameters - were activated at the thresholds set by the user, as indicated in the 'Technical Log'
IntelliSpace Corsium transmission | through study completion, an average of 1 year
  The Summary Record of Care (SRoC) data transmission from Tempus Pro to IntelliSpace Corsium will be independently reviewed for abnormalities and distortion by a clinician. The clinician will note any abnormalities altering diagnostic quality of the transmission.

OTHER OUTCOMES:
Adverse Device Effects | through study completion, an average of 1 year
  Frequency of Adverse Device Effects (ADE) related to device users - collected from Incident Reporting
Device Deficiencies | through study completion, an average of 1 year
  Frequency of Device Deficiencies (DD) - data collected from the technical data log recorded in the Tempus Pro at each Monitoring Event and from Product Complaint Reports

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lyon, MB CHB (HONS) MD MRCP FRCEM, Principal Investigator — CONSULTANT IN EMERGENCY MEDICINE, NHS LOTHIAN
Locations (1):
- Philips, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No